CLINICAL TRIAL: NCT03232853
Title: Evaluation of an E-learning to Prevent Drug Errors in Anesthesia.
Brief Title: E-learning to Prevent Drug Errors in Anesthesia
Acronym: ELPdrug
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0226
Record Dates: First submitted 2017-07-05; First posted 2017-07-28 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Medical Errors : Drugs Errors During Anesthesia
Keywords: medical error in anesthesia; drug error in anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Elearning — Elearning

SUMMARY:
The purpose of this observational study is to assess the efficiency of an e-learning in order to put into practice some preventive measures to avoid medication errors during anesthesia.

DETAILED DESCRIPTION:
Before the study, the investigators selected 15 preventive measures to avoid medication errors during anesthesia. These measures were learned to the entire anesthesia team (nurse, resident and anesthesiologist) during conventional meetings. An initial evaluation of the application of these measures will be carried out before the introduction of e-learning. This assessment will be conducted by nurses without the knowledge of the anesthetic team evaluated. After this initial evaluation, e-learning will be broadcast on the hospital intranet. Then a second evaluation of the application of the preventive measures will be carried out 6 month and 1 year after the introduction of e-learning.

ELIGIBILITY:
Inclusion criteria:

* patient undergoing regional and/or general anesthesia

Exclusion criteria:

* only sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing anesthesia in Lapeyronie Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of application of the preventive measures after versus before the use of an e-learning. | 1 day
  Percentage of application of the preventive measures after versus before the use of an e-learning.

SECONDARY OUTCOMES:
Evaluation of the application of each of the 15 preventive measureaccording to various clinical parameters | 1 day
  Evaluation of the application of each of the 15 preventive measures according to the clinical parameters of the patients followed (age of the patient, physical state of the ASA, type of surgery, type of anesthesia, period of the day or of the week, surgery of Emergency or elective.)emergency or elective surgery. In each completed questionnaire, these clinical parameters are noted.)

OTHER OUTCOMES:
Evaluation of the application of the preventive measures following the introduction of the e-learning in the anesthesia team. | 6 month and 1 year
  The evaluation of the application of the preventive measures will be assess following the introduction of the e-learning in the anesthesia team.

CONTACTS AND LOCATIONS:
Overall Officials: BIBOULET Philippe, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC